CLINICAL TRIAL: NCT06396702
Title: Emotion And Symptom-focused Engagement (EASE) Intervention for the Management of Emotional and Physical Symptoms Among Solid Organ Transplant Recipients-pilot Study
Brief Title: EASE-SOT Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Istvan Mucsi, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-6002
Record Dates: First submitted 2024-04-25; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Transplant;Failure,Kidney; Transplant; Failure, Heart; Transplant; Failure, Liver; Transplant; Failure, Pancreas; Transplant; Failure, Lung(S)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EASE-SOT Intervention Arm (Experimental): Participants in the intervention group receive EASE plus usual care. Each participant will participate in 8 EASE-psy sessions, starting twice a week during the inpatient stay and once every 1-2 weeks thereafter. They will also be screened for physical symptoms using electronic patient-reported outcome measures (ePROMs) twice a week while in-patient and once a week during the rest of the 8-week intervention period (EASE-phys). Participants will receive an output report that provides graphic representation of their current and previous scores on the various domains of health (e.g., depression, fatigue, etc.). If scoring above threshold for any symptom assessed during routine screening, participants will be referred/re-referred to a "symptom control" team. Additional ePROMs will be completed at baseline, 4, 8, 12 and 20 weeks.
  Interventions: Other: EASE-SOT
- Control Arm (No Intervention): Participants in the control group receive usual care alone. Additional ePROMs will be completed at baseline, 4, 8, 12 and 20 weeks.

INTERVENTIONS:
Other: EASE-SOT — EASE integrates supportive counseling and trauma-focused cognitive behavioral therapy (CBT) (EASE-psy) with systematic physical symptom screening and triggered referral to supportive care to manage moderate to severe physical symptoms (EASE-phys) using electronic patient reported outcome measures (ePROMs). The intervention duration is 8 weeks. Based on individual preference, EASE-psy may be administered in person or virtually via Microsoft Teams. Based on individual preference, participants may receive ePROMs either on tablets or to their personal electronic devices via email, while at the hospital ward and in clinics, ensuring easy access and administration of these tools.
  Arms: EASE-SOT Intervention Arm

SUMMARY:
Many transplant recipients may experience physical and emotional symptoms, such as anxiety, fatigue, sleep problems, pain, etc. Often, these symptoms are not reported or managed well, and can affect a patient's quality-of-life. Transplant recipients are grateful for the "gift of life" but physical and emotional symptoms reduce their quality-of-life. Transplant recipients and caregivers have felt unprepared for the ongoing symptoms and reduced quality-of-life post-transplant.

One way of monitoring and managing these symptoms is using the Emotion And Symptom-focused Engagement (EASE) intervention. EASE was originally developed for patients with acute leukemia and has begun to be adapted to help monitor and manage physical and emotional symptoms for organ transplant recipients.

EASE is comprised of two components:

1. Psychological - 8 supportive counselling sessions delivered by mental health clinicians to address concerns about mental health, losses from organ failure, coping with a transplant, experiences with living on the brink of death for a prolonged period of time, etc.
2. Physical - Regular assessments of physical symptoms using questionnaires and referral to healthcare professionals for symptom management as necessary.

EASE uses questionnaires, also called patient reported outcome measures (PROMs), for symptom assessment and monitoring. PROMs measure symptom severity, similarly to how bloodwork measures organ functioning. PROMs, as part of EASE, will ask recipients questions and help identify relevant physical, emotional, and social symptoms to enhance their care.

With the help of specialists, patients, and support from the Kidney Foundation of Canada, our team has begun to adapt the EASE intervention for transplant recipients. In order to finalize the adaptation of the EASE intervention for use in a routine transplant clinic, we are launching a pre-pilot study to gain real-life experience from managing symptoms of SOT recipients with the use of EASE-SOT.

DETAILED DESCRIPTION:
This is a parallel arm, randomized, controlled pilot study that will assess the feasibility for a large effectiveness trial using the EASE intervention to screen and manage emotional distress and physical symptoms among solid organ transplant (SOT) recipients. We will use a sequential cluster organization for recruitment. Initially, we will recruit kidney and kidney-pancreas transplant recipients, since we already have funding for this portion of our work. Subsequently, we will complete our study plan by recruiting liver, lung, and heart transplant recipients.

EASE integrates supportive counseling and trauma-focused cognitive behavioral therapy (CBT) (EASE-psy) with systematic physical symptom screening and triggered referral to supportive care to manage moderate to severe physical symptoms (EASE-phys). Participants in the intervention group receive EASE plus usual care. Each participant will participate in 8 EASE-psy sessions, starting twice a week during the inpatient stay and once every 1-2 week thereafter. They will also be screened for physical symptoms using electronic patient-reported outcome measures (ePROMs) twice a week while in-patient and once a week during the rest of the 8-week intervention period (EASE-phys).

Based on individual preference, participants will receive these ePROMs either on tablets or their personal electronic devices via email, while in the hospital ward or in clinics, ensuring easy access and administration of these tools. Participants will receive an output report that provides graphic representation of their current and previous scores on the various domains of health (e.g., depression, fatigue, etc.). This report will contain customized embedded URL links to the Symptomcare public domain. Embedded links will be in the form of: https://symptomcare.org/managing-my-symptoms-overview-patient/depression/?subjectid=1234&token=abcd. If scoring above threshold for any symptom assessed during routine screening, participants will be referred/re-referred to a "symptom control" team. Participants in the control group receive usual care alone. Additional ePROMs will be completed at baseline, 4, 8 12 and 20 weeks by patients in both arms.

ELIGIBILITY:
Inclusion Criteria:

* Participants consented pre-transplant: Potential transplant recipients who are listed on the waitlist and are identified by pre-transplant staff, recipients who have a living donor arranged (pertaining to kidney and liver recipients), participants currently completely pre-transplant prehabilitation (pertaining to lung and heart recipients), or those who are on the top of their respective organ transplant waitlists.
* Participants consented post-transplant: Incident kidney, kidney-pancreas, liver, lung, or heart transplant recipients identified during index transplant hospital admission at the inpatient transplant unit of the Ajmera Transplant Centre at Toronto General Hospital

Exclusion Criteria:

* Patients in ICU.
* Patients who are clinically unstable, have delirium or other severe mental health concern requiring psychiatric treatment - assessed by clinical team.
* Non-English speaking patients.
* Severe cognitive impairment as assessed by the recruitment and/or research team. This will be determined through communication with the organ transplant teams and by checking the patient's medical charts. If no cognitive impairment is indicated by the patients organ transplant team or is documented in their medical chart, the patient will be assessed to have no cognitive impairment.
* Unwilling or unable to provide informed consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Recruitment Target | Baseline
  Feasibility of the EASE-SOT intervention will be confirmed if our recruitment target of 120 participants (40 kidney and kidney-pancreas transplant recipients and 80 liver, lung, and heart transplant recipients) in a 30 month recruitment period is met.
Consent Rate | Baseline
  The consent rate describes the proportion of eligible patients who decline consent. Feasibility of the EASE-SOT intervention will be confirmed if the decline rate is ≤50%.
Retention Rate | Baseline to week 8 (8 weeks)
  The proportion of enrolled participants who continue to participate in the study at 8 weeks post-enrollment. Feasibility will be confirmed by a retention rate of 70%.
Adherence Rate | Baseline to week 20 (20 weeks)
  The proportion of enrolled participants who complete the EASE-Psy sessions, the symptom screening (EASE-phys) and outcome measures at the time offered, and have meetings the supportive care team if indicated by screens. Feasibility will be confirmed if ≥50% of participants complete EASE-psy sessions and symptom screening (EASE-phys) and outcome measures ≥50% of the time offered and have ≥1 meeting with the supportive care team if indicated by screens.
Drop-out Rate | Baseline to week 20 (20 weeks)
  The drop-out rate describes the proportion of enrolled participants who drop-out of the study for any reason (modality change, death, withdrawal, or loss to follow-up, etc.). Reasons for drop-out will be documented to assess the feasibility of the EASE-SOT intervention.
Patient Acceptability | Baseline to week 20 (20 weeks)
  Proportion of patients who find the EASE-SOT intervention 1) acceptable, 2) not burdensome, and 3) important based on responses to the "Patient Satisfaction Survey". Acceptability will be confirmed if >80% of patients find EASE acceptable.
Clinical Team Acceptability | Baseline to week 20 (20 weeks)
  Proportion of staff who find the EASE-SOT intervention intrusive to workflow, based on responses to the "Staff Satisfaction Survey". Acceptability will be confirmed if <20% of staff find the process intrusive to workflow.

SECONDARY OUTCOMES:
Incidence Rate of Healthcare Use | Baseline to week 20 (20 weeks)
  11-item recent healthcare use questions regarding healthcare use events such as recent hospitalizations, emergency visits, healthcare use. Incidence rates (event/100 patient years) of hospitalization, emergency admission, and hospitalization. Incidence rates will be compared between the two groups.
Post-transplant Quality of Life using the EQ-5D-5L | Baseline to week 20 (20 weeks)
  Measured by the the EuroQol-5 Dimension-5 Level (EQ5D5L) and Patient Reported Outcomes Measurement Information System (PROMIS) physical and mental health summary scores. The EQ5D5L measures quality of life (QOL) and utilities of health states by assessing mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a single item for each domain, measured on five response levels. We will use the Canadian value set. The PROMIS physical and mental health summary scores are calculated using responses to the domain specific item banks included in the PROMIS 29+2 v2.1 Profile measure.
Post-transplant Quality of Life using PROMIS physical and mental health summary scores | Baseline to week 20 (20 weeks)
  The Patient Reported Outcome Measurement Information System (PROMIS) 29+2 v1.2 profile assesses pain intensity using a single 0-10 numeric rating item, cognitive function using 2 items, and seven additional domains of health (physical function, fatigue, pain interference, depression, anxiety, ability to participate in social roles and activities, and sleep disturbance). The seven additional domains of health will be assessed using computer adaptive testing (CAT). The PROMIS 29 scales are scored on a T-score metric with a mean score of 50 and standard deviation of 10. For symptom domains, a higher score indicates a higher severity of that symptom. For function domains, a higher score indicates less impairment. The PROMIS physical and mental health summary scores are calculated using responses to the domain specific item banks included in the PROMIS 29+2 v2.1 Profile measure.
Presence of post-traumatic stress symptoms post-transplant using the SASRQ | Baseline to week 20 (20 weeks)
  Measured by the Stanford Acute Stress Reaction Questionnaire (SASRQ). The SASRQ is a 30-item questionnaire used to measure traumatic stress symptoms, including anxiety and dissociation symptoms, using a valid and reliable scale. The instructions were modified to refer to organ failure and the transplant surgery as the "traumatic event".
Presence of post-traumatic stress symptoms post-transplant using the PCL-5 | Baseline to week 20 (20 weeks)
  Measured by the Post-traumatic stress disorder checklist (PCL-5). The PCL-5 is a 20-item questionnaire used to measure traumatic stress using a valid and reliable scale. The self-report rating scale is 0-4 for each symptom, reflecting a change from 1-5 in the Diagnostic and Statistical Manual - IV (DSM-IV).
Severity of physical and emotional symptoms post-transplant | Baseline to week 20 (20 weeks)
  Measured by Patient Reported Outcomes Measurement Information System item banks administered using Computer Adaptive Testing (CAT) for anxiety, depression, dyspnea severity, fatigue, sleep disturbance, pain interference, pain intensity, physical function, cognitive function, and ability to participate in social roles and activities. For each domain specific item bank, responses to individual items are summed and converted into a standardized T-score, normalized to the US general population with a mean score of 50 and standard deviation of 10. For symptom domains, a higher score indicates a higher severity of that symptom. For function domains, a higher score indicates less impairment. When administered as CATs, 4 or more items are administered until standard error of measurement (SEM) is 0.30 or lower (equivalent to a reliability of 0.9 or higher) or 6 items have been asked. The recommended cut-off score for moderate-severe anxiety and depression symptoms on PROMIS tools is ≥60.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costanzo MR, Mills RM, Wynne J. Characteristics of "Stage D" heart failure: insights from the Acute Decompensated Heart Failure National Registry Longitudinal Module (ADHERE LM). Am Heart J. 2008 Feb;155(2):339-47. doi: 10.1016/j.ahj.2007.10.020. Epub 2007 Dec 19. PMID 18215606
- [Background] Ko DT, Alter DA, Austin PC, You JJ, Lee DS, Qiu F, Stukel TA, Tu JV. Life expectancy after an index hospitalization for patients with heart failure: a population-based study. Am Heart J. 2008 Feb;155(2):324-31. doi: 10.1016/j.ahj.2007.08.036. PMID 18215604
- [Background] Canadian Institute for Health Information, Canadian Organ Replacement Register annual report: treatment of end-stage organ failure in Canada, 2004 to 2013. 2015, Canadian Institute for Health Information: Ottawa, Ontario.
- [Background] Zelmer JL. The economic burden of end-stage renal disease in Canada. Kidney Int. 2007 Nov;72(9):1122-9. doi: 10.1038/sj.ki.5002459. Epub 2007 Aug 15. PMID 17700643
- [Background] ECONOMIC BURDEN OF ILLNESS IN CANADA, 2005-2008. 2017, Public Health Agency of Canada.
- [Background] Kidney Foundation of Canada, Facing the facts: includes highlights from the Canadian Organ Replacement Register. 2015.
- [Background] Klarenbach SW, Tonelli M, Chui B, Manns BJ. Economic evaluation of dialysis therapies. Nat Rev Nephrol. 2014 Nov;10(11):644-52. doi: 10.1038/nrneph.2014.145. Epub 2014 Aug 26. PMID 25157840
- [Background] Joshi VD. Quality of life in end stage renal disease patients. World J Nephrol. 2014 Nov 6;3(4):308-16. doi: 10.5527/wjn.v3.i4.308. PMID 25374827
- [Background] Tonelli M, Wiebe N, Knoll G, Bello A, Browne S, Jadhav D, Klarenbach S, Gill J. Systematic review: kidney transplantation compared with dialysis in clinically relevant outcomes. Am J Transplant. 2011 Oct;11(10):2093-109. doi: 10.1111/j.1600-6143.2011.03686.x. Epub 2011 Aug 30. PMID 21883901
- [Background] Molnar-Varga M, Molnar MZ, Szeifert L, Kovacs AZ, Kelemen A, Becze A, Laszlo G, Szentkiralyi A, Czira ME, Mucsi I, Novak M. Health-related quality of life and clinical outcomes in kidney transplant recipients. Am J Kidney Dis. 2011 Sep;58(3):444-52. doi: 10.1053/j.ajkd.2011.03.028. Epub 2011 Jun 12. PMID 21658828
- [Background] Kovacs AZ, Molnar MZ, Szeifert L, Ambrus C, Molnar-Varga M, Szentkiralyi A, Mucsi I, Novak M. Sleep disorders, depressive symptoms and health-related quality of life--a cross-sectional comparison between kidney transplant recipients and waitlisted patients on maintenance dialysis. Nephrol Dial Transplant. 2011 Mar;26(3):1058-65. doi: 10.1093/ndt/gfq476. Epub 2010 Aug 4. PMID 20685829
- [Background] CIHI, Annual Statistics on Organ Replacement in Canada: Dialysis, Transplantation and Donation, 2010 to 2019. 2020, Canadian Institute for Health Information: Ottawa, Ontario, Canada.
- [Background] Bryant RA, Creamer M, O'Donnell M, Silove D, McFarlane AC. The capacity of acute stress disorder to predict posttraumatic psychiatric disorders. J Psychiatr Res. 2012 Feb;46(2):168-73. doi: 10.1016/j.jpsychires.2011.10.007. Epub 2011 Nov 14. PMID 22088925
- [Background] Rosson S, Monaco F, Miola A, Cascino G, Stubbs B, Correll CU, Firth J, Ermis C, Perrotti A, Marciello F, Carvalho AF, Brunoni AR, Fusar-Poli P, Fornaro M, Gentile G, Granziol U, Pigato G, Favaro A, Solmi M. Longitudinal Course of Depressive, Anxiety, and Posttraumatic Stress Disorder Symptoms After Heart Surgery: A Meta-Analysis of 94 Studies. Psychosom Med. 2021 Jan 1;83(1):85-93. doi: 10.1097/PSY.0000000000000872. PMID 33021524
- [Background] Rodin G, Yuen D, Mischitelle A, Minden MD, Brandwein J, Schimmer A, Marmar C, Gagliese L, Lo C, Rydall A, Zimmermann C. Traumatic stress in acute leukemia. Psychooncology. 2013 Feb;22(2):299-307. doi: 10.1002/pon.2092. Epub 2011 Nov 13. PMID 22081505
- [Background] Zimmermann C, Yuen D, Mischitelle A, Minden MD, Brandwein JM, Schimmer A, Gagliese L, Lo C, Rydall A, Rodin G. Symptom burden and supportive care in patients with acute leukemia. Leuk Res. 2013 Jul;37(7):731-6. doi: 10.1016/j.leukres.2013.02.009. Epub 2013 Mar 11. PMID 23490030
- [Background] Nissim R, Zimmermann C, Minden M, Rydall A, Yuen D, Mischitelle A, Gagliese L, Schimmer A, Rodin G. Abducted by the illness: a qualitative study of traumatic stress in individuals with acute leukemia. Leuk Res. 2013 May;37(5):496-502. doi: 10.1016/j.leukres.2012.12.007. Epub 2013 Jan 24. PMID 23352641
- [Background] Rodin G, Deckert A, Tong E, Le LW, Rydall A, Schimmer A, Marmar CR, Lo C, Zimmermann C. Traumatic stress in patients with acute leukemia: A prospective cohort study. Psychooncology. 2018 Feb;27(2):515-523. doi: 10.1002/pon.4488. Epub 2017 Aug 10. PMID 28665521
- [Background] Szeifert L, Molnar MZ, Ambrus C, Koczy AB, Kovacs AZ, Vamos EP, Keszei A, Mucsi I, Novak M. Symptoms of depression in kidney transplant recipients: a cross-sectional study. Am J Kidney Dis. 2010 Jan;55(1):132-40. doi: 10.1053/j.ajkd.2009.09.022. Epub 2009 Nov 22. PMID 19932540
- [Background] Kwok, M., et al., Psychosocial distress and health related quality of life in kidney transplant recipients, in CST-CNTRP-SQT Joint Scientific Meeting 2017: Halifax, NS, Canada.
- [Background] Jin S, Xiang B, Zhong L, Yan L, Chen Z, Wang W, Xu M, Yang J. Quality of life and psychological distress of adult recipients after living donor liver transplantation. Transplant Proc. 2013 Jan-Feb;45(1):281-5. doi: 10.1016/j.transproceed.2012.05.076. PMID 23375316
- [Background] Baranyi A, Krauseneck T, Rothenhausler HB. Overall mental distress and health-related quality of life after solid-organ transplantation: results from a retrospective follow-up study. Health Qual Life Outcomes. 2013 Feb 8;11:15. doi: 10.1186/1477-7525-11-15. PMID 23391215
- [Background] Carbone M, Bufton S, Monaco A, Griffiths L, Jones DE, Neuberger JM. The effect of liver transplantation on fatigue in patients with primary biliary cirrhosis: a prospective study. J Hepatol. 2013 Sep;59(3):490-4. doi: 10.1016/j.jhep.2013.04.017. Epub 2013 Apr 27. PMID 23628322
- [Background] Kalaitzakis E, Josefsson A, Castedal M, Henfridsson P, Bengtsson M, Hugosson I, Andersson B, Bjornsson E. Factors related to fatigue in patients with cirrhosis before and after liver transplantation. Clin Gastroenterol Hepatol. 2012 Feb;10(2):174-81, 181.e1. doi: 10.1016/j.cgh.2011.07.029. Epub 2011 Aug 11. PMID 21839709
- [Background] McAdams-DeMarco MA, Olorundare IO, Ying H, Warsame F, Haugen CE, Hall R, Garonzik-Wang JM, Desai NM, Walston JD, Norman SP, Segev DL. Frailty and Postkidney Transplant Health-Related Quality of Life. Transplantation. 2018 Feb;102(2):291-299. doi: 10.1097/TP.0000000000001943. PMID 28885489
- [Background] Abbey SE, De Luca E, Mauthner OE, McKeever P, Shildrick M, Poole JM, Gewarges M, Ross HJ. Qualitative interviews vs standardized self-report questionnaires in assessing quality of life in heart transplant recipients. J Heart Lung Transplant. 2011 Aug;30(8):963-6. doi: 10.1016/j.healun.2011.03.017. Epub 2011 Apr 30. PMID 21531580
- [Background] Davison SN, Rathwell S, Ghosh S, George C, Pfister T, Dennett L. The Prevalence and Severity of Chronic Pain in Patients With Chronic Kidney Disease: A Systematic Review and Meta-Analysis. Can J Kidney Health Dis. 2021 Feb 19;8:2054358121993995. doi: 10.1177/2054358121993995. eCollection 2021. PMID 33680484
- [Background] Ju A, Unruh M, Davison SN, Dapueto J, Dew MA, Fluck R, Germain M, Jassal SV, Obrador G, O'Donoghue D, Howell M, O'Lone E, Shen JI, Craig JC, Tong A; SONG-HD Initiative. Identifying dimensions of fatigue in haemodialysis important to patients, caregivers and health professionals: An international survey. Nephrology (Carlton). 2020 Mar;25(3):239-247. doi: 10.1111/nep.13638. Epub 2019 Aug 16. PMID 31347227
- [Background] Pelgur H, Atak N, Kose K. Anxiety and depression levels of patients undergoing liver transplantation and their need for training. Transplant Proc. 2009 Jun;41(5):1743-8. doi: 10.1016/j.transproceed.2008.11.012. PMID 19545720
- [Background] Claxton RN, Blackhall L, Weisbord SD, Holley JL. Undertreatment of symptoms in patients on maintenance hemodialysis. J Pain Symptom Manage. 2010 Feb;39(2):211-8. doi: 10.1016/j.jpainsymman.2009.07.003. Epub 2009 Dec 5. PMID 19963337
- [Background] Barbera L, Sutradhar R, Howell D, Sussman J, Seow H, Dudgeon D, Atzema C, Earle C, Husain A, Liu Y, Krzyzanowska MK. Does routine symptom screening with ESAS decrease ED visits in breast cancer patients undergoing adjuvant chemotherapy? Support Care Cancer. 2015 Oct;23(10):3025-32. doi: 10.1007/s00520-015-2671-3. Epub 2015 Feb 26. PMID 25711657
- [Background] Di Maio M, Basch E, Bryce J, Perrone F. Patient-reported outcomes in the evaluation of toxicity of anticancer treatments. Nat Rev Clin Oncol. 2016 May;13(5):319-25. doi: 10.1038/nrclinonc.2015.222. Epub 2016 Jan 20. PMID 26787278
- [Background] Courtwright AM, Salomon S, Lehmann LS, Brettler T, Divo M, Camp P, Goldberg HJ, Wolfe DJ. The association between mood, anxiety and adjustment disorders and hospitalization following lung transplantation. Gen Hosp Psychiatry. 2016 Jul-Aug;41:1-5. doi: 10.1016/j.genhosppsych.2016.04.002. Epub 2016 Apr 28. PMID 27302717
- [Background] Ronksley PE, Hemmelgarn BR, Manns BJ, Wick J, James MT, Ravani P, Quinn RR, Scott-Douglas N, Lewanczuk R, Tonelli M. Potentially Preventable Hospitalization among Patients with CKD and High Inpatient Use. Clin J Am Soc Nephrol. 2016 Nov 7;11(11):2022-2031. doi: 10.2215/CJN.04690416. Epub 2016 Oct 6. PMID 27821636
- [Background] Basch E, Jia X, Heller G, Barz A, Sit L, Fruscione M, Appawu M, Iasonos A, Atkinson T, Goldfarb S, Culkin A, Kris MG, Schrag D. Adverse symptom event reporting by patients vs clinicians: relationships with clinical outcomes. J Natl Cancer Inst. 2009 Dec 2;101(23):1624-32. doi: 10.1093/jnci/djp386. Epub 2009 Nov 17. PMID 19920223
- [Background] Jensen RE, Snyder CF, Abernethy AP, Basch E, Potosky AL, Roberts AC, Loeffler DR, Reeve BB. Review of electronic patient-reported outcomes systems used in cancer clinical care. J Oncol Pract. 2014 Jul;10(4):e215-22. doi: 10.1200/JOP.2013.001067. Epub 2013 Dec 3. PMID 24301843
- [Background] Stover AM, Basch EM. Using patient-reported outcome measures as quality indicators in routine cancer care. Cancer. 2016 Feb 1;122(3):355-7. doi: 10.1002/cncr.29768. Epub 2015 Nov 30. No abstract available. PMID 26619153
- [Background] Basch E. Patient-Reported Outcomes - Harnessing Patients' Voices to Improve Clinical Care. N Engl J Med. 2017 Jan 12;376(2):105-108. doi: 10.1056/NEJMp1611252. No abstract available. PMID 28076708
- [Background] Basch E, Deal AM, Dueck AC, Scher HI, Kris MG, Hudis C, Schrag D. Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment. JAMA. 2017 Jul 11;318(2):197-198. doi: 10.1001/jama.2017.7156. PMID 28586821
- [Background] Rodrigue JR, Nelson DR, Hanto DW, Reed AI, Curry MP. Patient-reported immunosuppression nonadherence 6 to 24 months after liver transplant: association with pretransplant psychosocial factors and perceptions of health status change. Prog Transplant. 2013 Dec;23(4):319-28. doi: 10.7182/pit2013501. PMID 24311395
- [Background] Scholz U, Klaghofer R, Dux R, Roellin M, Boehler A, Muellhaupt B, Noll G, Wuthrich RP, Goetzmann L. Predicting intentions and adherence behavior in the context of organ transplantation: gender differences of provided social support. J Psychosom Res. 2012 Mar;72(3):214-9. doi: 10.1016/j.jpsychores.2011.10.008. Epub 2012 Jan 5. PMID 22325701
- [Background] Morales JM, Varo E, Lazaro P. Immunosuppressant treatment adherence, barriers to adherence and quality of life in renal and liver transplant recipients in Spain. Clin Transplant. 2012 Mar-Apr;26(2):369-76. doi: 10.1111/j.1399-0012.2011.01544.x. Epub 2011 Oct 30. PMID 22035067
- [Background] Burra P, Germani G, Gnoato F, Lazzaro S, Russo FP, Cillo U, Senzolo M. Adherence in liver transplant recipients. Liver Transpl. 2011 Jul;17(7):760-70. doi: 10.1002/lt.22294. PMID 21384527
- [Background] Dobbels F, Vanhaecke J, Dupont L, Nevens F, Verleden G, Pirenne J, De Geest S. Pretransplant predictors of posttransplant adherence and clinical outcome: an evidence base for pretransplant psychosocial screening. Transplantation. 2009 May 27;87(10):1497-504. doi: 10.1097/TP.0b013e3181a440ae. PMID 19461486
- [Background] Dew MA, Dabbs AD, Myaskovsky L, Shyu S, Shellmer DA, DiMartini AF, Steel J, Unruh M, Switzer GE, Shapiro R, Greenhouse JB. Meta-analysis of medical regimen adherence outcomes in pediatric solid organ transplantation. Transplantation. 2009 Sep 15;88(5):736-46. doi: 10.1097/TP.0b013e3181b2a0e0. PMID 19741474
- [Background] Chisholm-Burns MA, Spivey CA, Wilks SE. Social support and immunosuppressant therapy adherence among adult renal transplant recipients. Clin Transplant. 2010 May-Jun;24(3):312-20. doi: 10.1111/j.1399-0012.2009.01060.x. Epub 2009 Aug 19. PMID 19694770
- [Background] Fredericks EM, Lopez MJ, Magee JC, Shieck V, Opipari-Arrigan L. Psychological functioning, nonadherence and health outcomes after pediatric liver transplantation. Am J Transplant. 2007 Aug;7(8):1974-83. doi: 10.1111/j.1600-6143.2007.01878.x. PMID 17617862
- [Background] Akman B, Uyar M, Afsar B, Sezer S, Ozdemir FN, Haberal M. Adherence, depression and quality of life in patients on a renal transplantation waiting list. Transpl Int. 2007 Aug;20(8):682-7. doi: 10.1111/j.1432-2277.2007.00495.x. Epub 2007 May 29. PMID 17535307
- [Background] Penkower L, Dew MA, Ellis D, Sereika SM, Kitutu JM, Shapiro R. Psychological distress and adherence to the medical regimen among adolescent renal transplant recipients. Am J Transplant. 2003 Nov;3(11):1418-25. doi: 10.1046/j.1600-6135.2003.00226.x. PMID 14525604
- [Background] Wiebe C, Nevins TE, Robiner WN, Thomas W, Matas AJ, Nickerson PW. The Synergistic Effect of Class II HLA Epitope-Mismatch and Nonadherence on Acute Rejection and Graft Survival. Am J Transplant. 2015 Aug;15(8):2197-202. doi: 10.1111/ajt.13341. Epub 2015 Jun 11. PMID 26095765
- [Background] Tielen M, van Exel J, Laging M, Beck DK, Khemai R, van Gelder T, Betjes MG, Weimar W, Massey EK. Attitudes to medication after kidney transplantation and their association with medication adherence and graft survival: a 2-year follow-up study. J Transplant. 2014;2014:675301. doi: 10.1155/2014/675301. Epub 2014 Apr 28. PMID 24868449
- [Background] Epstein AS, Goldberg GR, Meier DE. Palliative care and hematologic oncology: the promise of collaboration. Blood Rev. 2012 Nov;26(6):233-9. doi: 10.1016/j.blre.2012.07.001. Epub 2012 Aug 5. PMID 22874874
- [Background] Engel GL. The need for a new medical model: a challenge for biomedicine. Science. 1977 Apr 8;196(4286):129-36. doi: 10.1126/science.847460.
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Davison SN. Patient-Oriented Research: Clinical Innovation Based on CKD Patients' Priorities for Care. Am J Kidney Dis. 2016 Dec;68(6):833-835. doi: 10.1053/j.ajkd.2016.09.004. No abstract available. PMID 27884279
- [Background] Davison SN, Jassal SV. Supportive Care: Integration of Patient-Centered Kidney Care to Manage Symptoms and Geriatric Syndromes. Clin J Am Soc Nephrol. 2016 Oct 7;11(10):1882-1891. doi: 10.2215/CJN.01050116. Epub 2016 Aug 10. PMID 27510454
- [Background] Li M, Macedo A, Crawford S, Bagha S, Leung YW, Zimmermann C, Fitzgerald B, Wyatt M, Stuart-McEwan T, Rodin G. Easier Said Than Done: Keys to Successful Implementation of the Distress Assessment and Response Tool (DART) Program. J Oncol Pract. 2016 May;12(5):e513-26. doi: 10.1200/JOP.2015.010066. Epub 2016 Apr 5. PMID 27048610
- [Background] Zimmermann C, Pope A, Hannon B, Krzyzanowska MK, Rodin G, Li M, Howell D, Knox JJ, Leighl NB, Sridhar S, Oza AM, Prince R, Lheureux S, Hansen AR, Rydall A, Chow B, Herx L, Booth CM, Dudgeon D, Dhani N, Liu G, Bedard PL, Mathews J, Swami N, Le LW. Phase II Trial of Symptom Screening With Targeted Early Palliative Care for Patients With Advanced Cancer. J Natl Compr Canc Netw. 2021 Sep 7;20(4):361-370.e3. doi: 10.6004/jnccn.2020.7803. PMID 34492632
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Rodin G, An E, Shnall J, Malfitano C. Psychological Interventions for Patients With Advanced Disease: Implications for Oncology and Palliative Care. J Clin Oncol. 2020 Mar 20;38(9):885-904. doi: 10.1200/JCO.19.00058. Epub 2020 Feb 5. PMID 32023159
- [Background] Barrett, T.A., Outpatient Cardiac Palliative Care Reduces Healthcare Utilization. The Journal of Heart and Lung Transplantation, 2020. 39(4, Supplement): p. S362.
- [Background] Colman R, Singer LG, Barua R, Downar J. Characteristics, interventions, and outcomes of lung transplant recipients co-managed with palliative care. J Palliat Med. 2015 Mar;18(3):266-9. doi: 10.1089/jpm.2014.0167. Epub 2014 Aug 27. PMID 25162457
- [Background] Baumann AJ, Wheeler DS, James M, Turner R, Siegel A, Navarro VJ. Benefit of Early Palliative Care Intervention in End-Stage Liver Disease Patients Awaiting Liver Transplantation. J Pain Symptom Manage. 2015 Dec;50(6):882-6.e2. doi: 10.1016/j.jpainsymman.2015.07.014. Epub 2015 Aug 22. PMID 26303186
- [Background] Freeman N, Le LW, Singer LG, Colman R, Zimmermann C, Wentlandt K. Impact of a transplant palliative care clinic on symptoms for patients awaiting lung transplantation. J Heart Lung Transplant. 2016 Aug;35(8):1037-9. doi: 10.1016/j.healun.2016.05.006. Epub 2016 May 16. No abstract available. PMID 27311372
- [Background] Pullen LC. Bringing palliative care to transplant. Am J Transplant. 2021 Jul;21(7):2315-2316. doi: 10.1111/ajt.16035. No abstract available. PMID 34196485
- [Background] Wentlandt K, Dall'Osto A, Freeman N, Le LW, Kaya E, Ross H, Singer LG, Abbey S, Clarke H, Zimmermann C. The Transplant Palliative Care Clinic: An early palliative care model for patients in a transplant program. Clin Transplant. 2016 Dec;30(12):1591-1596. doi: 10.1111/ctr.12838. Epub 2016 Nov 4. PMID 27910190
- [Background] Denis F, Lethrosne C, Pourel N, Molinier O, Pointreau Y, Domont J, Bourgeois H, Senellart H, Tremolieres P, Lizee T, Bennouna J, Urban T, El Khouri C, Charron A, Septans AL, Balavoine M, Landry S, Solal-Celigny P, Letellier C. Randomized Trial Comparing a Web-Mediated Follow-up With Routine Surveillance in Lung Cancer Patients. J Natl Cancer Inst. 2017 Sep 1;109(9). doi: 10.1093/jnci/djx029. PMID 28423407
- [Background] Gheihman G, Zimmermann C, Deckert A, Fitzgerald P, Mischitelle A, Rydall A, Schimmer A, Gagliese L, Lo C, Rodin G. Depression and hopelessness in patients with acute leukemia: the psychological impact of an acute and life-threatening disorder. Psychooncology. 2016 Aug;25(8):979-89. doi: 10.1002/pon.3940. Epub 2015 Sep 18. PMID 26383625
- [Background] Rodin G, Malfitano C, Rydall A, Schimmer A, Marmar CM, Mah K, Lo C, Nissim R, Zimmermann C. Emotion And Symptom-focused Engagement (EASE): a randomized phase II trial of an integrated psychological and palliative care intervention for patients with acute leukemia. Support Care Cancer. 2020 Jan;28(1):163-176. doi: 10.1007/s00520-019-04723-2. Epub 2019 Apr 17. PMID 31001692
- [Background] Bansal, A., et al., Accuracy of the PROMIS-57 Depression and Anxiety Scales in Kidney Transplant Recipients, in CST-CNTRP-SQT Joint Scientific Meeting. 2017: Halifax, NS, Canada.
- [Background] Tang, E., et al. Validation of the PROMIS-57 and PROMIS-29 short form profile questionnaires in patients undergoing Hemodialysis. in Annual General Meeting of the Canadian Society of Nephrology. 2018. Vancouver, BC.
- [Background] Tang E, Bansal A, Novak M, Mucsi I. Patient-Reported Outcomes in Patients with Chronic Kidney Disease and Kidney Transplant-Part 1. Front Med (Lausanne). 2018 Jan 15;4:254. doi: 10.3389/fmed.2017.00254. eCollection 2017. PMID 29379784
- [Background] Tang E, Ekundayo O, Peipert JD, Edwards N, Bansal A, Richardson C, Bartlett SJ, Howell D, Li M, Cella D, Novak M, Mucsi I. Validation of the Patient-Reported Outcomes Measurement Information System (PROMIS)-57 and -29 item short forms among kidney transplant recipients. Qual Life Res. 2019 Mar;28(3):815-827. doi: 10.1007/s11136-018-2058-2. Epub 2018 Nov 22. PMID 30467780
- [Background] Wong D, Cao S, Ford H, Richardson C, Belenko D, Tang E, Ugenti L, Warsmann E, Sissons A, Kulandaivelu Y, Edwards N, Novak M, Li M, Mucsi I. Exploring the use of tablet computer-based electronic data capture system to assess patient reported measures among patients with chronic kidney disease: a pilot study. BMC Nephrol. 2017 Dec 6;18(1):356. doi: 10.1186/s12882-017-0771-7. PMID 29212466
- [Background] Cardena E, Koopman C, Classen C, Waelde LC, Spiegel D. Psychometric properties of the Stanford Acute Stress Reaction Questionnaire (SASRQ): a valid and reliable measure of acute stress. J Trauma Stress. 2000 Oct;13(4):719-34. doi: 10.1023/A:1007822603186. PMID 11109242
- [Background] Fries JF, Cella D, Rose M, Krishnan E, Bruce B. Progress in assessing physical function in arthritis: PROMIS short forms and computerized adaptive testing. J Rheumatol. 2009 Sep;36(9):2061-6. doi: 10.3899/jrheum.090358. PMID 19738214
- [Background] Papuga MO, Dasilva C, McIntyre A, Mitten D, Kates S, Baumhauer JF. Large-scale clinical implementation of PROMIS computer adaptive testing with direct incorporation into the electronic medical record. Health Syst (Basingstoke). 2017 Dec 7;7(1):1-12. doi: 10.1057/s41306-016-0016-1. eCollection 2018. PMID 31214335
- [Background] Segawa E, Schalet B, Cella D. A comparison of computer adaptive tests (CATs) and short forms in terms of accuracy and number of items administrated using PROMIS profile. Qual Life Res. 2020 Jan;29(1):213-221. doi: 10.1007/s11136-019-02312-8. Epub 2019 Oct 8. PMID 31595451
- [Background] Smith AB, Hanbury A, Retzler J. Item banking and computer-adaptive testing in clinical trials: Standing in sight of the PROMISed land. Contemp Clin Trials Commun. 2018 Nov 17;13:005-5. doi: 10.1016/j.conctc.2018.11.005. eCollection 2019 Mar. PMID 30582066
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- [Background] Hays RD, Spritzer KL, Schalet BD, Cella D. PROMIS(R)-29 v2.0 profile physical and mental health summary scores. Qual Life Res. 2018 Jul;27(7):1885-1891. doi: 10.1007/s11136-018-1842-3. Epub 2018 Mar 22. PMID 29569016
- [Background] Li B, Cairns JA, Draper H, Dudley C, Forsythe JL, Johnson RJ, Metcalfe W, Oniscu GC, Ravanan R, Robb ML, Roderick P, Tomson CR, Watson CJE, Bradley JA. Estimating Health-State Utility Values in Kidney Transplant Recipients and Waiting-List Patients Using the EQ-5D-5L. Value Health. 2017 Jul-Aug;20(7):976-984. doi: 10.1016/j.jval.2017.01.011. Epub 2017 May 12. PMID 28712628
- [Background] Sayah FA, Bansback N, Bryan S, Ohinmaa A, Poissant L, Pullenayegum E, Xie F, Johnson JA. Determinants of time trade-off valuations for EQ-5D-5L health states: data from the Canadian EQ-5D-5L valuation study. Qual Life Res. 2016 Jul;25(7):1679-85. doi: 10.1007/s11136-015-1203-4. Epub 2015 Dec 10. PMID 26659899
- [Background] Xie F, Pullenayegum E, Gaebel K, Bansback N, Bryan S, Ohinmaa A, Poissant L, Johnson JA; Canadian EQ-5D-5L Valuation Study Group. A Time Trade-off-derived Value Set of the EQ-5D-5L for Canada. Med Care. 2016 Jan;54(1):98-105. doi: 10.1097/MLR.0000000000000447. PMID 26492214
- [Background] Tang E, Dano S, Edwards N, Macanovic S, Ford H, Bartlett S, Howell D, Li M, Novak M, Mucsi I. Screening for symptoms of anxiety and depression in patients treated with renal replacement therapy: utility of the Edmonton Symptom Assessment System-Revised. Qual Life Res. 2022 Feb;31(2):597-605. doi: 10.1007/s11136-021-02910-5. Epub 2021 Jun 17. PMID 34138450
- [Background] Dano S, Pokarowski M, Liao B, Tang E, Ekundayo O, Li V, Edwards N, Ford H, Novak M, Mucsi I. Evaluating symptom burden in kidney transplant recipients: validation of the revised Edmonton Symptom Assessment System for kidney transplant recipients - a single-center, cross-sectional study. Transpl Int. 2020 Apr;33(4):423-436. doi: 10.1111/tri.13572. Epub 2020 Jan 30. PMID 31919903
- [Background] Report, T.-H.T., We ask because we care- The Tri-Hospital + TPH Health Equity Data Collection Research Project Report. 2013: p. 51.
- [Background] Taylor K, Chu NM, Chen X, Shi Z, Rosello E, Kunwar S, Butz P, Norman SP, Crews DC, Greenberg KI, Mathur A, Segev DL, Shafi T, McAdams-DeMarco MA. Kidney Disease Symptoms before and after Kidney Transplantation. Clin J Am Soc Nephrol. 2021 Jul;16(7):1083-1093. doi: 10.2215/CJN.19031220. Epub 2021 Jun 18. PMID 34597266
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Bovin MJ, Marx BP, Weathers FW, Gallagher MW, Rodriguez P, Schnurr PP, Keane TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in veterans. Psychol Assess. 2016 Nov;28(11):1379-1391. doi: 10.1037/pas0000254. Epub 2015 Dec 14. PMID 26653052
- [Background] Butler LD, Koopman C, Classen C, Spiegel D. Traumatic stress, life events, and emotional support in women with metastatic breast cancer: cancer-related traumatic stress symptoms associated with past and current stressors. Health Psychol. 1999 Nov;18(6):555-60. doi: 10.1037//0278-6133.18.6.555. PMID 10619528
- [Background] Koopman C, Gore-Felton C, Azimi N, O'Shea K, Ashton E, Power R, De Maria S, Israelski D, Spiegel D. Acute stress reactions to recent life events among women and men living with HIV/AIDS. Int J Psychiatry Med. 2002;32(4):361-78. doi: 10.2190/CK2N-33NV-3PVF-GLVR. PMID 12779186
- [Background] Koopman C, Gore-Felton C, Classen C, Kim P, Spiegel D. Acute stress reactions to everyday stressful life events among sexual abuse survivors with PTSD. J Child Sex Abus. 2001;10(2):83-99. doi: 10.1300/j070v10n02_05. PMID 15149937
- [Background] Rodin, G. and L.A. Gillies, Individual Psychotherapy for the Patient with Advanced Disease, in Handbook of Psychiatry in Palliative Medicine, W.B. Harvey Max Chochinov, Editor. 2009, Oxford University Press: New York. p. 189-196.
- [Background] Marmar, C. and C. Henn-Haase, Anxiety Reduction Treatment for Acute Trauma (ARTAT): Treatment Manual. . 2011, New York, NY: New York University.
- [Background] Rodin G, Lo C, Rydall A, Shnall J, Malfitano C, Chiu A, Panday T, Watt S, An E, Nissim R, Li M, Zimmermann C, Hales S. Managing Cancer and Living Meaningfully (CALM): A Randomized Controlled Trial of a Psychological Intervention for Patients With Advanced Cancer. J Clin Oncol. 2018 Aug 10;36(23):2422-2432. doi: 10.1200/JCO.2017.77.1097. Epub 2018 Jun 29. PMID 29958037
- [Background] Spiegel, D. and P. Spira, Supportive-Expressive Group Therapy: A Treatment Manual of Psychosocial Intervention for Women with Recurrent Breast Cancer. 1991, Stanford, CA: Psychosocial Treatment Laboratory, Stanford University School of Medicine.
- [Background] Perepletchikova, F. and A.E. Kazdin, Treatment Integrity and Therapeutic Change: Issues and Research Recommendations. Clinical Psychology: Science and Practice, 2005. 12(4): p. 365-383.
- [Background] Bruera E, Kuehn N, Miller MJ, Selmser P, Macmillan K. The Edmonton Symptom Assessment System (ESAS): a simple method for the assessment of palliative care patients. J Palliat Care. 1991 Summer;7(2):6-9. PMID 1714502
- [Background] Hannon B, Swami N, Pope A, Rodin G, Dougherty E, Mak E, Banerjee S, Bryson J, Ridley J, Zimmermann C. The oncology palliative care clinic at the Princess Margaret Cancer Centre: an early intervention model for patients with advanced cancer. Support Care Cancer. 2015 Apr;23(4):1073-80. doi: 10.1007/s00520-014-2460-4. Epub 2014 Oct 4. PMID 25281230
- [Background] Ontario, C.C., Symptom Management Guides to Practice. Website accessed October 11, 2020.
- [Background] Zimmermann C, Swami N, Krzyzanowska M, Hannon B, Leighl N, Oza A, Moore M, Rydall A, Rodin G, Tannock I, Donner A, Lo C. Early palliative care for patients with advanced cancer: a cluster-randomised controlled trial. Lancet. 2014 May 17;383(9930):1721-30. doi: 10.1016/S0140-6736(13)62416-2. Epub 2014 Feb 19. PMID 24559581
- [Background] Lee RT, Ramchandran K, Sanft T, Von Roenn J. Implementation of supportive care and best supportive care interventions in clinical trials enrolling patients with cancerdagger. Ann Oncol. 2015 Sep;26(9):1838-1845. doi: 10.1093/annonc/mdv207. Epub 2015 Apr 28. PMID 25922064
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Teare MD, Dimairo M, Shephard N, Hayman A, Whitehead A, Walters SJ. Sample size requirements to estimate key design parameters from external pilot randomised controlled trials: a simulation study. Trials. 2014 Jul 3;15:264. doi: 10.1186/1745-6215-15-264. PMID 24993581
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476